CLINICAL TRIAL: NCT00962598
Title: The Role Of Omega-3 Fatty Acids In Adolescent Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Vilma Gabbay, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 12-1321; R21AT004576-01 (NIH)
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Depressive Disorder, Major
Keywords: Adolescents; Major Depressive Disorder; Proton Magnetic Resonance Spectroscopy; Immune System Activation; Omega-3 Fatty Acids
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fatty Acids, Omega-3; Fish Oils; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Corn Oil (Placebo Comparator): The dosage will correspond to the titration schedule of the Omega-3 Fatty Acid experimental treatment.
  Interventions: Dietary Supplement: Corn oil
- Omega-3 Fatty Acids (Experimental): The initial dose will be 1.2g/d. This will be increased gradually by 0.6 per 2 weeks to a possible maximum daily dose of 3.6 g/d.
  Interventions: Drug: Omega 3 Fatty Acids

INTERVENTIONS:
Drug: Omega 3 Fatty Acids — The study medication will consist of combined EPA/DHA with a ratio of 2:1. Dosage will be titrated based on clinical response and side effects. The initial dose will be 1.2g/d. This will be increased gradually by 0.6 per 2 weeks to a possible maximum daily dose of 3.6 g/d. Patients will have to remain on a dose for 2 weeks to provide the opportunity to assess clinical response at any one dose. The total duration of the intervention will be 10 weeks.
  Other Names: Fish oil
  Arms: Omega-3 Fatty Acids
Dietary Supplement: Corn oil — The dosage will correspond to the titration schedule of the Omega-3 Fatty Acid experimental treatment. Placebo (corn oil) and omega-3FA capsules will be identical in color and smell.
  Arms: Corn Oil

SUMMARY:
The purpose of this study is to examine the effects of a 10-week Omega-3 Fatty Acid treatment phase on brain chemistry of adolescents with major depressive disorder (MDD) using proton magnetic resonance imaging.

DETAILED DESCRIPTION:
This study rests on a confluence of findings showing that: 1) Major depressive disorder (MDD), is a major public health concern that often emerges in adolescence; which entails 2) pathophysiological abnormalities in fronto-striatal structures resulting in death and atrophy of glia and neurons; 3) omega-3 fatty acids (FA) effects on brain function in adolescent MDD can be assessed by proton magnetic resonance spectroscopy (1H MRS); and, 4) it is critical that commonly used complementary and alternative medicines such as omega-3FA that have face validity be tested for their neurobiological effect in MDD.

Using 1H MRSI, this study examines the effects of Omega-3FA on striatal and anterior cingulate cortex (ACC) concentrations of the neurocellular biomarkers total choline (tCho), total creatine (tCr), and γ-aminobutyric acid (GABA, ACC only) in adolescent MDD. Hypotheses are: 1) relative to placebo, omega-3FA treatment will result in significant reductions of striatal and ACC tCho and tCr concentrations, and increased ACC GABA; 2: Regardless of treatment condition (placebo or Omega-3FA), MDD adolescents who are improved at the end of 10-week treatment will exhibit a significant decrease in striatal and ACC tCho and tCr concentrations, and increases in ACC GABA relative to unimproved adolescents.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 19 years old (inclusive) of both sexes and all ethnic/racial groups.
* DSM-IV-TR criteria for MDD
* MDD Duration of at least 8 weeks and a severity score of at least 40 on the CDRS-R.
* Age at first onset MDD of at least 12 years.
* No significant medical or neurological disorder
* For female subjects, negative pregnancy test at time of enrollment.
* Female subjects who are sexually active and not using a method of birth control will be excluded. Use of hormonal contraceptives (such as prescribed "birth control pills" or a prescribed birth control implant) is not exclusionary.
* Subjects must be able to swallow capsules.
* A minimum IQ of 80 will be required.

Exclusion Criteria:

* Current or Past DSM-IV-TR diagnoses of bipolar disorder, schizophrenia, psychosis, autism/pervasive developmental disorder (PDD), and Tourette's disorder (TD).
* Current diagnosis of eating disorder, panic disorder, obsessive-compulsive disorder (OCD), post traumatic stress disorder (PTSD), conduct disorder, and substance related disorders other than nicotine.
* Current suicidal ideation with intent or plan, or who may pose a danger to themselves.
* Current antidepressant treatment will be excluded. Past antidepressant treatment will not be exclusionary, so long as patients are off antidepressant medication for 60 days prior to study entry. No individual will be advised to terminate ongoing treatment.
* Certain short half-life medications, such as vitamins that contain unidentified ingredients, St. Johns Wort, S-adenosyl Methionine (SAM), clonidine, and some over-the-counter medications.
* A minimum of 90 days off of treatment with long half life medications, such as neuroleptics, prior to study entry is required. Stimulant medication treatment for ADHD will not be exclusionary.
* If adolescents have been in psychotherapy prior to their entry in the study, they will be allowed to continue with the treatment. However, psychotherapy cannot be initiated at the time of study entry.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Gabbay, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Gabbay V, Freed RD, Alonso CM, Senger S, Stadterman J, Davison BA, Klein RG. A Double-Blind Placebo-Controlled Trial of Omega-3 Fatty Acids as a Monotherapy for Adolescent Depression. J Clin Psychiatry. 2018 Jun 26;79(4):17m11596. doi: 10.4088/JCP.17m11596. PMID 29985566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in December 2005, with enrollment from January 2006 to June 2013. Participants recruited for this imaging from another study, GCO 12-1321.
Groups:
- Corn Oil: Corn oil: The dosage correspond to the titration schedule of the Omega-3 Fatty Acid experimental treatment. Placebo (corn oil) and omega-3FA capsules will be identical in color and smell.
Period: Overall Study
Arm/Group | Corn Oil | Omega-3 Fatty Acids
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corn Oil | Omega-3 Fatty Acids | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.62 (3.087) | 16.51 (2.756) | 16.56 (2.805)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: ACC Glx/Water
Description: The data reflects the ratio of Glutamine-Glutamate and water in the brain (ratio divided by 10000 for analysis purposes). Glutamate is a precursor to Glutamine, an amino acid which functions as an excitatory neurotransmitter in the human brain.
Time Frame: baseline and 10-weeks
Measure: Mean (Standard Deviation); unit: ratio * 10^-4
Arm/Group | Corn Oil | Omega-3 Fatty Acids
Number analyzed (Participants) | 7 | 9
ratio * 10^-4
  ACC Glx/Water Baseline | 19.21 (5.173) | 18.99 (2.989)
  ACC Glx/Water 10 weeks | 19.28 (3.339) | 20.61 (5.201)

2. Primary Outcome: ACC GABA/Water
Description: The ratio of gamma-Aminobutyric acid (GABA) and water in the brain (ratio divided by 10000 for analysis purposes), that was observed in MR Spectroscopy. GABA, an amino acid produced by cells of the central nervous system, is an inhibitory neurotransmitter, prominent in the human brain.
Time Frame: baseline and 10-weeks
Measure: Mean (Standard Deviation); unit: ratio * 10^-4
Arm/Group | Corn Oil | Omega-3 Fatty Acids
Number analyzed (Participants) | 7 | 9
ratio * 10^-4
  ACC GABA/Water Baseline | 28.37 (4.097) | 25.28 (2.845)
  ACC GABA/Water 10 weeks | 28.93 (5.200) | 28.84 (3.512)

ADVERSE EVENTS:
Arm/Group | Corn Oil | Omega-3 Fatty Acids
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes